CLINICAL TRIAL: NCT05763017
Title: A Randomized Comparative Trial of Relative Motion Splint Versus Metacarpophalangeal Joint Blocking Splint in the Management of Trigger Finger
Brief Title: Comparing Relative Motion Splint and Metacarpophalangeal Joint Blocking Splint for Trigger Finger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JEP-2022-319
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Trigger Finger; Stenosing Tenosynovitis
Keywords: relative motion splint; metacarpophalangeal joint blocking splint
MeSH Terms: conditions — Trigger Finger Disorder; Tendon Entrapment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relative Motion Splint (Experimental): In the relative motion splint, the metacarpophalangeal joint of the affected finger(s) positioned in approximately 20°-25° more extension/flexion than metacarpophalangeal joint of the adjacent fingers.
  Interventions: Other: Relative Motion Splint
- Metacarpophalangeal Joint Blocking Splint (Active Comparator): In the metacarpophalangeal joint blocking splint, the metacarpophalangeal joint of the affected finger(s) positioned in 0°.
  Interventions: Other: Metacarpophalangeal Joint Blocking Splint

INTERVENTIONS:
Other: Relative Motion Splint — Six weeks relative motion splint wear.
  Arms: Relative Motion Splint
Other: Metacarpophalangeal Joint Blocking Splint — Six weeks metacarpophalangeal joint blocking splint wear.
  Arms: Metacarpophalangeal Joint Blocking Splint

SUMMARY:
The purpose of this study is to compare the effectiveness of relative motion splint and metacarpophalangeal joint blocking splints in terms of sign and symptoms, hand function, occupational performance, and perception of splint wearability (comfort and satisfaction) after six weeks of TF management.

ELIGIBILITY:
Inclusion Criteria:

* single or multiple trigger finger
* unilateral or bilateral trigger finger
* neutral metacarpophalangeal joint position can be attained during passive isolated metacarpophalangeal joint extension of the affected finger

Exclusion Criteria:

* trigger thumb
* steroid injection of the affected finger within last six months
* A1 pulley release of the affected finger.
* history of fracture, tendon injury, nerve injury, Dupuytren's contracture, and other soft tissue injuries of the affected finger or adjacent fingers.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Stages of Stenosing Tenosynovitis (SST) | Baseline, 6 weeks after splint wear
  SST is a grading system that divides trigger finger into six stages. Stage 1 is normal; Stage 2 is uneven finger movement; Stage 3 is triggering or clicking or catching; Stage 4 is locking of finger in flexion or extension, which can be unlocked by active finger movement; Stage 5 is locking of finger in flexion or extension, which requires application of passive force to unlock; and Stage 6 is locked finger in flexion or extension

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for pain | Baseline, 6 weeks after splint wear
  The left end of the VAS labelled as "no pain" and the right end labelled as "extreme pain".
Number of triggering events in ten active fists | Baseline, 6 weeks after splint wear
  The number of triggering events (0 - 10) can be obtained by asking the patient to make 10 active full fists.
Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure | Baseline, 6 weeks after splint wear
  DASH is a 30-item, self-report questionnaire that range from 0-100 score, with higher scores represent more severe disability or poorer hand function.
Canadian Occupational Performance Measure (COPM) | Baseline, 6 weeks after splint wear
  COPM is a interview-based assessment tool for measuring occupational performance. The importance, satisfaction, and performance of an activity are rated using a 10-point rating scale.
Visual Analog Scale (VAS) for splint comfort | Baseline, 3 and 6 weeks after splint wear
  The left end of the VAS labelled as "not at all comfortable' and the right end labelled as "extremely comfortable".
Visual Analog Scale (VAS) for splint satisfaction | Baseline, 3 and 6 weeks after splint wear
  The left end of the VAS labelled as "not at all satisfied" and the right end labelled as "extremely satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Siaw Chui Chai, PhD (OT), Principal Investigator — Occupational Therapy Programme, Center for Rehabilitation & Special Needs Studies (iCaRehab)
Locations (1):
- Hospital Sultan Haji Ahmad Shah, Temerluh, Pahang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leong LX, Chai SC, Howell JW, Rasdi HFM, Rahman NRA. A randomized comparative trial: Relative motion vs metacarpophalangeal joint blocking orthoses for trigger finger management. J Hand Ther. 2025 Jul 4:S0894-1130(25)00090-0. doi: 10.1016/j.jht.2025.05.018. Online ahead of print. PMID 40617791
- [Derived] Leong LX, Chai SC, Howell JW, Mohd Rasdi HF, Abdul Rahman NR. Relative motion splints versus metacarpophalangeal joint blocking splints in the management of trigger finger: Study protocol for a randomized comparative trial. PLoS One. 2024 Aug 13;19(8):e0307033. doi: 10.1371/journal.pone.0307033. eCollection 2024. PMID 39137205